CLINICAL TRIAL: NCT04640311
Title: A Two-part, Randomized, Double-blind, Single-dose, Crossover Study to Compare Formulations Produced by Two Methods of Manufacture for Bioequivalence and Dissolution in Healthy Adult Volunteers
Brief Title: Comparison of Daprodustat Formulations Produced by Two Methods of Manufacture for Bioequivalence and Dissolution in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 213022
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Anaemia
Keywords: Daprodustat; Pharmacokinetic; Bioequivalence; Bioavailability
MeSH Terms: conditions — Anemia | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Daprodustat Dissolution 1/Dissolution 2/Reference (Experimental)
  Interventions: Drug: Daprodustat
- Part A: Daprodustat Dissolution 2/Reference/Dissolution 1 (Experimental)
  Interventions: Drug: Daprodustat
- Part A: Daprodustat Reference/Dissolution 1/Dissolution 2 (Experimental)
  Interventions: Drug: Daprodustat
- Part B: Daprodustat Process 1/ Process 2 (Experimental)
  Interventions: Drug: Daprodustat
- Part B: Daprodustat Process 2/ Process 1 (Experimental)
  Interventions: Drug: Daprodustat

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be available as oral tablets.

SUMMARY:
This study is comprised of two discrete Parts. Part A is a 3-period cross over evaluating relative bioavailability. Part B is a 2-period cross over evaluating bioequivalence. There will be a minimum of a 7-day washout period between treatment periods. Participants will participate in Part A or Part B, but not both. Approximately 200 participants will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants must be overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests. A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator and/or the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Participants with body weight more than or equal to (>=) 45 kilogram (kg) and body mass index (BMI) within the range 19-31 kg per meter square (Kg/m^2).
* Male or female
* A female participant is eligible to participate if she is not breastfeeding, and at least; not pregnant as confirmed by pregnancy testing or not a woman of childbearing potential (WOCBP) or agrees to follow the contraceptive guidance during the treatment period to the follow-up visit.
* Participants capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants with history of malignancy within the prior 2 years or currently receiving treatment for cancer. The only exception is localized squamous- or basal-cell carcinoma of the skin definitively treated 12 weeks or more prior to enrolment.
* Participants unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 30 days prior to Day 1 in this study. Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation (administration of last dose of investigational study treatment) within the last 30 days (or 5 half-lives, whichever is longer) before Day 1 in this study in any other clinical study involving an investigational study intervention or any other type of medical research.
* Part A participants may not participate in Part B, and Part B participants may not participate in Part A if enrolment is concurrent or overlaps.
* Participants with positive pre-study drug/alcohol screen.
* Participants with regular use of known drugs of abuse.
* Participants with a positive laboratory confirmation of Coronavirus disease 2019 (COVID-19) infection, or high clinical index of suspicion for COVID-19.
* Participants with regular alcohol consumption within 6 months prior to the study.
* Participants with urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine containing products (nicotine patches or vaporizing devices) within 6 months prior to screening.
* Participants with sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Shaddinger B, Mahar KM, Sprys M, Andrews SM, Chattoraj S, Israni R, Cobitz A. Comparison of Two Manufacturing Processes of Daprodustat for Bioequivalence and Dissolution in Healthy Volunteers: A Randomized Crossover Study. Clin Pharmacol Drug Dev. 2023 Jul;12(7):739-748. doi: 10.1002/cpdd.1257. Epub 2023 May 1. PMID 37125459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across 4 centers in the United States. This study consisted of two parts; Part A (3-period crossover study) and Part B (2-period crossover study).
Pre-assignment Details: A total of 259 participants (52 in Part A and 207 in Part B) were enrolled in the study (Safety Population: It comprised of all randomized participants who have taken at least 1 dose of study intervention).
Groups:
- Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1: Participants received a single oral dose of daprodustat 4 milligrams (mg) tablets with dissolution profile (DP) 1 made by Process 2 (high shear wet granulation) in Treatment Period 1 followed by a single oral dose of daprodustat 4 mg tablets with DP 2 made by Process 2 in Treatment Period 2. Participants were administered a single oral dose of daprodustat 4 mg tablets made by reference Process 1 (twin screw granulation) in Treatment Period 3. There was a washout of at least 7 days after daprodustat dosing in Treatment Periods 1 and 2. Participants were followed up for 7 days after last dose in Treatment Period 3.
- Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2: Participants received a single oral dose of daprodustat 4 mg tablets with DP 2 made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 4 mg tablets made by reference Process 1 in Treatment Period 2. Participants were administered a single oral dose of daprodustat 4 mg tablets with DP 1 made by Process 2 in Treatment Period 3. There was a washout of at least 7 days after daprodustat dosing in Treatment Periods 1 and 2. Participants were followed up for 7 days after last dose in Treatment Period 3.
- Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2: Participants received a single oral dose of daprodustat 4 mg tablets made by reference Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 4 mg tablets with DP 1 made by Process 2 in Treatment Period 2. Participants were administered a single oral dose of daprodustat 4 mg tablets with DP 2 made by Process 2 in Treatment Period 3. There was a washout of at least 7 days after daprodustat dosing in Treatment Periods 1 and 2. Participants were followed up for 7 days after last dose in Treatment Period 3.
- Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1: Participants received a single oral dose of daprodustat 1 mg tablets made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 1 mg tablets made by Process 1 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2: Participants received a single oral dose of daprodustat 1 mg tablets made by Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 1 mg tablets made by Process 2 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1: Participants received a single oral dose of daprodustat 2 mg tablets made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 2 mg tablets made by Process 1 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2: Participants received a single oral dose of daprodustat 2 mg tablets made by Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 2 mg tablets made by Process 2 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1: Participants received a single oral dose of daprodustat 4 mg tablets made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 4 mg tablets made by Process 1 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2: Participants received a single oral dose of daprodustat 4 mg tablets made by Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 4 mg tablets made by Process 2 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1: Participants received a single oral dose of daprodustat 6 mg tablets made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 6 mg tablets made by Process 1 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2: Participants received a single oral dose of daprodustat 6 mg tablets made by Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 6 mg tablets made by Process 2 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1: Participants received a single oral dose of daprodustat 8 mg tablets made by Process 2 in Treatment Period 1 followed by a single oral dose of daprodustat 8 mg tablets made by Process 1 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
- Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2: Participants received a single oral dose of daprodustat 8 mg tablets made by Process 1 in Treatment Period 1 followed by a single oral dose of daprodustat 8 mg tablets made by Process 2 in Treatment Period 2. There was a washout of at least 7 days after daprodustat dosing in Treatment Period 1. Participants were followed up for 7 days after last dose in Treatment Period 2.
Period: Part A:Treatment Period 1 (Up to 2 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 16 | 18 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 16 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn by sponsor due to impact of inclement weather events | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Washout 1 (Up to 7 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 15 | 16 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 15 | 16 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A:Treatment Period 2 (Up to 2 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 15 | 16 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn by sponsor due to impact of inclement weather events | 3 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Washout 2 (Up to 7 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 12 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A:Treatment Period 3 (Up to 2 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 12 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B:Treatment Period 1 (Up to 2 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 0 | 0 | 0 | 21 | 19 | 21 | 22 | 21 | 21 | 21 | 21 | 20 | 20
Completed | 0 | 0 | 0 | 20 | 19 | 20 | 20 | 21 | 19 | 21 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part B: Washout 1 (Up to 7 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 0 | 0 | 0 | 20 | 19 | 20 | 20 | 21 | 19 | 21 | 20 | 20 | 20
Completed | 0 | 0 | 0 | 20 | 19 | 20 | 20 | 21 | 19 | 21 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Treatment Period 2(Up to 2 Days)
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2
Started | 0 | 0 | 0 | 20 | 19 | 20 | 20 | 21 | 19 | 21 | 20 | 20 | 20
Completed | 0 | 0 | 0 | 20 | 19 | 20 | 20 | 21 | 19 | 21 | 20 | 19 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were presented for Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Daprodustat DP 1 Process 2/Daprodustat DP 2 Process 2/Daprodustat Process 1 | Part A: Daprodustat DP 2 Process 2/ Daprodustat Process 1 / Daprodustat DP 1 Process 2 | Part A: Daprodustat Process 1 / Daprodustat DP 1 Process 2/ Daprodustat DP 2 Process 2 | Part B: Daprodustat 1 mg Process 2/ Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 1/Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 2/Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 1/ Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 2/ Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 1/Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 2/Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 1/Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 2/Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 1/Daprodustat 8 mg Process 2 | Total
Number analyzed (Participants) | 16 | 18 | 18 | 21 | 19 | 21 | 22 | 21 | 21 | 21 | 21 | 20 | 20 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 18 | 21 | 19 | 21 | 22 | 21 | 21 | 21 | 21 | 20 | 20 | 259
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 8 | 7 | 11 | 10 | 4 | 8 | 6 | 4 | 5 | 4 | 86
  Male | 11 | 12 | 10 | 13 | 12 | 10 | 12 | 17 | 13 | 15 | 17 | 15 | 16 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 9
  Black or African American | 4 | 4 | 7 | 8 | 10 | 9 | 9 | 11 | 13 | 5 | 2 | 12 | 17 | 111
  Mixed Race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  White - Arabic/ North African Heritage | 1 | 3 | 1 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 12
  White - White/ Caucasian/ European Heritage | 10 | 10 | 9 | 8 | 3 | 5 | 6 | 9 | 3 | 13 | 14 | 7 | 3 | 100
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Asian - Central/ South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Asian - East Asian Heritage | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
  Asian - Japanese Heritage | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 9
  Asian - Mixed Race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Concentration-time Curve (AUC) From Zero (Pre-dose) to Time of Last Quantifiable Concentration (AUC[0-t]) Following Administration of Daprodustat
Description: Blood samples were collected at indicated time points to investigate the pharmacokinetics of daprodustat. Pharmacokinetic analysis was conducted using standard non-compartmental methods. The geometric coefficient of variation is model adjusted and is a within-participant coefficient of variation. Analysis was performed using a mixed effect model.
Time Frame: Pre-dose and 30 minutes, 1 Hour, 2 Hours, 2 Hours 30 Minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours Post-dose in Treatment Periods 1, 2 and 3
Population: Pharmacokinetic Population comprised of all participants in the Safety Population (All randomized participants who have taken at least 1 dose of study intervention) who had at least 1 non-missing Pharmacokinetic assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Groups:
- Part A: Daprodustat Process 1: Participants received a single oral dose of daprodustat 4 mg tablets made by reference Process 1 in each of the Treatment Periods 1, 2 and 3.
- Part A: Daprodustat Process 2 Dissolution Profile 1: Participants received a single oral dose of daprodustat 4 mg tablets with dissolution profile 1 made by Process 2 in each of the Treatment Periods 1, 2 and 3.
- Part A: Daprodustat Process 2 Dissolution Profile 2: Participants received a single oral dose of daprodustat 4 mg tablets with dissolution profile 2 made by Process 2 in each of the Treatment Periods 1, 2 and 3.
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 35 | 35 | 34
Hours*nanograms per milliliter | 155.5 (14.7) | 159.9 (14.7) | 158.5 (14.7)
Statistical Analysis 1: Comparison: Part A: Daprodustat Process 1 vs Part A: Daprodustat Process 2 Dissolution Profile 1; Test type: Other; Geometric mean ratio = 1.028, 90% CI 2-sided [0.9699 to 1.090] — Geometric mean ratio of Daprodustat Process 1 to Process 2 Dissolution Profile 1 has been presented
Statistical Analysis 2: Comparison: Part A: Daprodustat Process 1 vs Part A: Daprodustat Process 2 Dissolution Profile 2; Test type: Other; Geometric mean ratio = 1.019, 90% CI 2-sided [0.9602 to 1.081] — Geometric mean ratio of Daprodustat Process 1 to Process 2 Dissolution Profile 2 has been presented

2. Primary Outcome: Part B: AUC(0-t) Following Administration of Daprodustat
Description: as for outcome 1
Time Frame: Pre-dose and 30 minutes, 1 Hour, 2 Hours, 2 Hours 30 Minutes, 3 Hours, 4 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours Post-dose in Treatment Periods 1 and 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Groups:
- Part B: Daprodustat 1 mg Process 1: Participants received a single oral dose of daprodustat 1 mg tablets made by Process 1 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 1 mg Process 2: Participants received a single oral dose of daprodustat 1 mg tablets made by Process 2 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 2 mg Process 1: Participants received a single oral dose of daprodustat 2 mg tablets made by Process 1 in each of the Treatment Periods 1 and 2
- Part B: Daprodustat 2 mg Process 2: Participants received a single oral dose of daprodustat 2 mg tablets made by Process 2 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 4 mg Process 1: Participants received a single oral dose of daprodustat 4 mg tablets made by Process 1 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 4 mg Process 2: Participants received a single oral dose of daprodustat 4 mg tablets made by Process 2 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 6 mg Process 1: Participants received a single oral dose of daprodustat 6 mg tablets made by Process 1 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 6 mg Process 2: Participants received a single oral dose of daprodustat 6 mg tablets made by Process 2 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 8 mg Process 1: Participants received a single oral dose of daprodustat 8 mg tablets made by Process 1 in each of the Treatment Periods 1 and 2.
- Part B: Daprodustat 8 mg Process 2: Participants received a single oral dose of daprodustat 8 mg tablets made by Process 2 in each of the Treatment Periods 1 and 2.
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 39 | 40 | 42 | 41 | 42 | 40 | 42 | 41 | 40 | 40
Hours*nanograms per milliliter | 36.97 (13.5) | 38.02 (13.5) | 83.27 (17.0) | 79.08 (17.0) | 132.9 (15.4) | 134.2 (15.4) | 249.5 (16.3) | 241.5 (16.3) | 292.8 (16.3) | 278.5 (16.3)
Statistical Analysis 1: Comparison: Part B: Daprodustat 1 mg Process 1 vs Part B: Daprodustat 1 mg Process 2; Test type: Equivalence — Bioequivalence was to be determined if the 90 percent (%) confidence interval (CI) of ratio's of geometric means (geometric mean of Process 2/Process 1) falls within a range of 0.80 to 1.25; Geometric mean ratio = 1.029, 90% CI 2-sided [0.9770 to 1.083] — Geometric mean ratio of Daprodustat 1 mg Process 2 to Process 1 has been presented
Statistical Analysis 2: Comparison: Part B: Daprodustat 2 mg Process 1 vs Part B: Daprodustat 2 mg Process 2; Test type: Equivalence — Bioequivalence was to be determined if the 90% CI of ratio's of geometric means (geometric mean of Process 2/Process 1) falls within a range of 0.80 to 1.25; Geometric mean ratio = 0.9496, 90% CI 2-sided [0.8914 to 1.012] — Geometric mean ratio of Daprodustat 2 mg Process 2 to Process 1 has been presented
Statistical Analysis 3: Comparison: Part B: Daprodustat 4 mg Process 1 vs Part B: Daprodustat 4 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 1.010, 90% CI 2-sided [0.9533 to 1.070] — Geometric mean ratio of Daprodustat 4 mg Process 2 to Process 1 has been presented
Statistical Analysis 4: Comparison: Part B: Daprodustat 6 mg Process 1 vs Part B: Daprodustat 6 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9679, 90% CI 2-sided [0.9115 to 1.028] — Geometric mean ratio of Daprodustat 6 mg Process 2 to Process 1 has been presented
Statistical Analysis 5: Comparison: Part B: Daprodustat 8 mg Process 1 vs Part B: Daprodustat 8 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9511, 90% CI 2-sided [0.8948 to 1.011] — Geometric mean ratio of Daprodustat 8 mg Process 2 to Process 1 has been presented

3. Primary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) Following Administration of Daprodustat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 35 | 35 | 34
Nanograms per milliliter | 68.22 (28.7) | 71.06 (28.7) | 71.51 (28.7)
Statistical Analysis 1: Comparison: Part A: Daprodustat Process 1 vs Part A: Daprodustat Process 2 Dissolution Profile 1; Test type: Other; Geometric mean ratio = 1.042, 90% CI 2-sided [0.9308 to 1.166] — Geometric mean ratio of Daprodustat Process 1 to Process 2 Dissolution Profile 1 has been presented
Statistical Analysis 2: Comparison: Part A: Daprodustat Process 1 vs Part A: Daprodustat Process 2 Dissolution Profile 2; Test type: Other; Geometric mean ratio = 1.048, 90% CI 2-sided [0.9349 to 1.175] — Geometric mean ratio of Daprodustat Process 1 to Process 2 Dissolution Profile 2 has been presented

4. Primary Outcome: Part B: Cmax Following Administration of Daprodustat
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 39 | 40 | 42 | 41 | 42 | 40 | 42 | 41 | 40 | 40
Nanograms per milliliter | 17.90 (22.2) | 17.39 (22.2) | 39.20 (28.8) | 35.30 (28.8) | 62.05 (30.9) | 60.21 (30.9) | 113.4 (26.7) | 109.7 (26.7) | 139.5 (27.6) | 120.0 (27.6)
Statistical Analysis 1: Comparison: Part B: Daprodustat 1 mg Process 1 vs Part B: Daprodustat 1 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9716, 90% CI 2-sided [0.8936 to 1.056] — Geometric mean ratio of Daprodustat 1 mg Process 2 to Process 1 has been presented
Statistical Analysis 2: Comparison: Part B: Daprodustat 2 mg Process 1 vs Part B: Daprodustat 2 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9006, 90% CI 2-sided [0.8107 to 1.000] — Geometric mean ratio of Daprodustat 2 mg Process 2 to Process 1 has been presented
Statistical Analysis 3: Comparison: Part B: Daprodustat 4 mg Process 1 vs Part B: Daprodustat 4 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9703, 90% CI 2-sided [0.8665 to 1.087] — Geometric mean ratio of Daprodustat 4 mg Process 2 to Process 1 has been presented
Statistical Analysis 4: Comparison: Part B: Daprodustat 6 mg Process 1 vs Part B: Daprodustat 6 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.9675, 90% CI 2-sided [0.8778 to 1.066] — Geometric mean ratio of Daprodustat 6 mg Process 2 to Process 1 has been presented
Statistical Analysis 5: Comparison: Part B: Daprodustat 8 mg Process 1 vs Part B: Daprodustat 8 mg Process 2; Test type: Equivalence — [test comment as in outcome 2, analysis 2]; Geometric mean ratio = 0.8606, 90% CI 2-sided [0.7770 to 0.9532] — Geometric mean ratio of Daprodustat 8 mg Process 2 to Process 1 has been presented

5. Secondary Outcome: Part A: AUC From Zero Time (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) Following Administration of Daprodustat
Description: Blood samples were collected at indicated time points to investigate the pharmacokinetics of daprodustat. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanograms per milliliter
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 34 | 35 | 33
Hours* nanograms per milliliter | 159.9 (34.7) | 162.5 (31.5) | 161.5 (34.7)

6. Secondary Outcome: Part A: Time of Occurrence of Cmax (Tmax) Following Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 35 | 35 | 34
Hours | 2.500 [0.500 to 8.00] | 2.000 [1.00 to 6.00] | 2.000 [1.00 to 4.00]

7. Secondary Outcome: Part A: Terminal Phase Half-life (T1/2) Following Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 34 | 35 | 33
Hours | 1.797 (28.9) | 1.910 (25.0) | 1.932 (34.0)

8. Secondary Outcome: Part A: Apparent Clearance Following Oral Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 34 | 35 | 33
Liters per hour | 25.02 (34.7) | 24.61 (31.5) | 24.77 (34.7)

9. Secondary Outcome: Part A: Apparent Volume of Distribution Following Oral Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2
Number analyzed (Participants) | 34 | 35 | 33
Liters | 64.87 (42.4) | 67.81 (47.3) | 69.05 (50.9)

10. Secondary Outcome: Part B: AUC(0-inf) Following Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanograms per milliliter
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 36 | 37 | 42 | 41 | 40 | 39 | 42 | 40 | 39 | 39
Hours* nanograms per milliliter | 37.71 (33.1) | 38.81 (37.8) | 84.36 (36.0) | 78.59 (34.1) | 135.5 (32.7) | 135.2 (33.0) | 250.4 (38.7) | 246.0 (40.5) | 295.8 (38.5) | 282.7 (39.3)

11. Secondary Outcome: Part B: Tmax Following Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 39 | 40 | 42 | 41 | 42 | 40 | 42 | 41 | 40 | 40
Hours | 2.000 [0.500 to 4.00] | 2.000 [0.517 to 4.00] | 2.250 [1.00 to 4.00] | 2.000 [0.500 to 4.00] | 2.000 [1.00 to 4.00] | 2.000 [0.500 to 4.00] | 2.000 [0.500 to 4.00] | 1.000 [0.500 to 4.00] | 2.000 [1.00 to 4.00] | 2.000 [0.500 to 6.00]

12. Secondary Outcome: Part B: T1/2 Following Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 36 | 37 | 42 | 41 | 40 | 39 | 42 | 40 | 39 | 39
Hours | 1.162 (28.2) | 1.163 (30.2) | 1.545 (32.3) | 1.489 (32.6) | 1.814 (31.2) | 1.775 (26.5) | 1.852 (24.5) | 1.920 (24.4) | 1.997 (35.3) | 2.136 (35.0)

13. Secondary Outcome: Part B: Apparent Clearance Following Oral Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 36 | 37 | 42 | 41 | 40 | 39 | 42 | 40 | 39 | 39
Liters per hour | 26.52 (33.1) | 25.76 (37.8) | 23.71 (36.0) | 25.45 (34.1) | 29.53 (32.7) | 29.58 (33.0) | 23.96 (38.7) | 24.39 (40.5) | 27.04 (38.5) | 28.30 (39.3)

14. Secondary Outcome: Part B: Apparent Volume of Distribution Following Oral Administration of Daprodustat
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
Number analyzed (Participants) | 36 | 37 | 42 | 41 | 40 | 39 | 42 | 40 | 39 | 39
Liters | 44.45 (31.7) | 43.22 (43.6) | 52.83 (43.1) | 54.65 (30.9) | 77.28 (43.9) | 75.74 (40.3) | 64.02 (37.1) | 67.56 (38.9) | 77.92 (54.5) | 87.21 (42.6)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (non-SAEs) were collected up to 27 days in Part A and up to 18 days in Part B of the study.
Description: Safety Population was used to assess all-cause mortality, SAEs and non-SAEs which comprised of all randomized participants who have taken at least 1 dose of study intervention. AEs were presented part-wise and treatment-wise.
Arm/Group | Part A: Daprodustat Process 1 | Part A: Daprodustat Process 2 Dissolution Profile 1 | Part A: Daprodustat Process 2 Dissolution Profile 2 | Part B: Daprodustat 1 mg Process 1 | Part B: Daprodustat 1 mg Process 2 | Part B: Daprodustat 2 mg Process 1 | Part B: Daprodustat 2 mg Process 2 | Part B: Daprodustat 4 mg Process 1 | Part B: Daprodustat 4 mg Process 2 | Part B: Daprodustat 6 mg Process 1 | Part B: Daprodustat 6 mg Process 2 | Part B: Daprodustat 8 mg Process 1 | Part B: Daprodustat 8 mg Process 2
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/43 | 0/39 | 0/40 | 0/42 | 0/41 | 0/42 | 0/40 | 0/42 | 0/41 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/43 | 0/39 | 0/40 | 0/42 | 0/41 | 1/42 | 0/40 | 0/42 | 0/41 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/46 | 3/45 | 0/43 | 1/39 | 1/40 | 3/42 | 1/41 | 3/42 | 5/40 | 6/42 | 1/41 | 5/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Daprodustat Process 1 (N=46) | Part A: Daprodustat Process 2 Dissolution Profile 1 (N=45) | Part A: Daprodustat Process 2 Dissolution Profile 2 (N=43) | Part B: Daprodustat 1 mg Process 1 (N=39) | Part B: Daprodustat 1 mg Process 2 (N=40) | Part B: Daprodustat 2 mg Process 1 (N=42) | Part B: Daprodustat 2 mg Process 2 (N=41) | Part B: Daprodustat 4 mg Process 1 (N=42) | Part B: Daprodustat 4 mg Process 2 (N=40) | Part B: Daprodustat 6 mg Process 1 (N=42) | Part B: Daprodustat 6 mg Process 2 (N=41) | Part B: Daprodustat 8 mg Process 1 (N=40) | Part B: Daprodustat 8 mg Process 2 (N=40)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Daprodustat Process 1 (N=46) | Part A: Daprodustat Process 2 Dissolution Profile 1 (N=45) | Part A: Daprodustat Process 2 Dissolution Profile 2 (N=43) | Part B: Daprodustat 1 mg Process 1 (N=39) | Part B: Daprodustat 1 mg Process 2 (N=40) | Part B: Daprodustat 2 mg Process 1 (N=42) | Part B: Daprodustat 2 mg Process 2 (N=41) | Part B: Daprodustat 4 mg Process 1 (N=42) | Part B: Daprodustat 4 mg Process 2 (N=40) | Part B: Daprodustat 6 mg Process 1 (N=42) | Part B: Daprodustat 6 mg Process 2 (N=41) | Part B: Daprodustat 8 mg Process 1 (N=40) | Part B: Daprodustat 8 mg Process 2 (N=40)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04640311/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04640311/SAP_001.pdf